CLINICAL TRIAL: NCT03537378
Title: A Multi-Center Clinical Study of the Hybrid APC Therapy in Early Central Lung Neoplasms
Brief Title: Hybrid APC Therapy in Early Central Lung Neoplasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiayuan Sun (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director,Endoscopy Department,Shanghai Chest Hospital Affiliation: Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHCHE201801
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Lung Neoplasms
Keywords: Hybrid APC,Early Central Lung Neoplasms,
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hybrid APC Therapy Group (Experimental): 1) Patients are diagnosed as early central lung neoplasms (severe dysplasia, carcinoma in situ, microinvasive carcinoma，mucoepidermoid carcinoma.etc.) by inquiry of the first doctor, CT test, endoscopy and histopathology. Patients who meet inclusion/exclusion criteria are not suitable for or refuse surgery.
  Interventions: Procedure: Hybrid APC

INTERVENTIONS:
Procedure: Hybrid APC — • HybridAPC is integrated with traditional APC and water-jet technique, which has been successfully applied for endoscopic treatment of mucosal lesions in GI, such as Barrett esophageal and lesions in colon. Submucosal injection of water jet can elevate superficial lesion, and then APC can be more effective in ablation of superficial tumor with a protection for muscular layer. The application of HybridAPC in respiratory intervention could theoretically protect cartilage, adventitia, reduce damage and formation of scare, and increase ablation energy to reach radical treatment. • High-frequency EBUS, could display the boundary between cartilage endomembrane and cartilage, in order to determine the depth of tumor.

SUMMARY:
1.1 Aims：This cohort study aims to investigate the clinical value of Hybrid APC for treatment of early central lung neoplasms.

1.2 methods：A total of 30 patients with early central lung neoplasms will be included in this open, multicenter, prospective study. Primary observation endpoint is recorded at 3 months follow-up, and after 3 months patients could be continued to follow up. The data are expressed in terms of mean and percentage. The categorical variables are analyzed by chi-square test, and the four table data is analyzed using the exact probability method. The continuous variable analysis is used by t test. Statistical analysis is performed with SPSS 20.0 software. P < 0.05 is considered statistically significant.

DETAILED DESCRIPTION:
This is a prospective, multicenter, and cohort study. Study subjects: patients with early central lung neoplasms meet inclusion/exclusion criteria and could receive interventional therapy.

There are 3 study site in this study and a total of 30 patients with early central lung cancer will be included.

HybridAPC is integrated with traditional APC and water-jet technique, which has been successfully applied for endoscopic treatment of mucosal lesions in GI, such as Barrett esophageal and lesions in colon. Submucosal injection of water jet can elevate superficial lesion, and then APC can be more effective in ablation of superficial tumor with a protection for muscular layer. The application of HybridAPC in respiratory intervention could theoretically protect cartilage, adventitia, reduce damage and formation of scare, and increase ablation energy to reach radical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Bronchoscopy and fluorescence bronchoscopy found endoluminal growth lesions of upper segmental bronchus. AFB indicates malignant possibility.
2. Size ≤ 20 mm
3. Flat, nodule or polypoid type
4. Negative imaging: HRCT indicates no tumor in lung and lymph node enlargement; or PET-CT finds no lesions in lung or suspicious lymph node tumors involve.
5. Clinical stage: Tis or T1N0M0
6. High-grade intraepithelial neoplasia (including severe atypical dysplasia and carcinoma in situ) mucoepidermoid carcinomaand ,squamous cancer and etc. confirmed by biopsy histopathology
7. High-frequency EBUS indicates the depth of lesions is cartilage endomembrane or internal part of adventitia of tracheal membranous part
8. Patients are not suitable for surgery or refuse surgery
9. Inform consent is available

Exclusion Criteria:

1. Patients with severe cardiopulmonary dysfunction or other contraindication can not tolerate endoscopic examination and treatment
2. Severe bleeding tendency
3. Poor compliance
4. Unstable vital signs
5. Investigators consider subjects should not be included because of specific situations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Successful remission rate: | 3 months
  successful remission is defined as absence of intraepithelial neoplasia in biopsies of original locations at 3 months after HybridAPC upon follow up

SECONDARY OUTCOMES:
Complications | 3 months
  possible complications include perforation, bleeding, fever, stenosis, cough and etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided